CLINICAL TRIAL: NCT02220959
Title: Is Preoperative Exercise Test in Morbid Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy a Predictive Test for Extubation?
Brief Title: Is Preoperative Exercise Test in Morbid Obese Patients a Predictive Test for Extubation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, professor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 14467
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Morbid Obesity
Keywords: morbid obesity surgery; walk test; exercise
MeSH Terms: conditions — Obesity, Morbid; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- walk test (Experimental): morbid obese patients (BMI>40) undergoing laparoscopic sleeve gastrectomy walking 60 meters under 1 minute before and after the measurement of Forced vital capacity (FVC)
  Interventions: Other: walk test

INTERVENTIONS:
Other: walk test — patients will be encouraged to walk a 60 meter distance under 1 minute and FVC will be measured before and after the walk test
  Other Names: 60 meter walk test

SUMMARY:
the purpose of this study is to determine if 60 meter test done prior to surgery is a predictive in terms of extubation in morbid obese patients undergoing morbid obese surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients between 18-60 years old
* patients with BMI > 40
* patients undergoing Laparoscopic Sleeve Gastrectomy

Exclusion Criteria:

* patients with Chronic obstructive pulmonary disease (COPD), Asthma,
* patients with uncompensated heart failure
* Uncompensated diabetes mellitus
* Patients Who have orthopedic problems that effects the exercise test

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with successful extubation | postoperative 30 minutes
  preoperative 60 meter walk test

CONTACTS AND LOCATIONS:
Locations (1):
- Cerrahpasa medical Faculty General surgery operation theatre, Istanbul, Turkey (Türkiye)